CLINICAL TRIAL: NCT01346228
Title: USING SMART PHONE TECHNOLOGY AS A PLATFORM FOR DELIVERING MENTAL HEALTH CARE TO RURAL VETERANS
Brief Title: Using Smart Phone Technology To Rural Veterans
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Collaborators: South Central VA Mental Illness Research, Education & Clinical Center (U.S. Federal Agency)
Responsible Party: Ellen Teng, PhD., Michael E. DeBakey VA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-28199
Record Dates: First submitted 2011-04-29; First posted 2011-05-02 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2011-04

CONDITIONS: Panic Disorders; Anxiety Disorders
Keywords: Panic; Panic Disorder; Anxiety
MeSH Terms: conditions — Panic Disorder; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Panic Control Treatment (PCT) — 2 Day treatment for Panic Disorder
  Other Names: Panic Group; Weekend Panic Group

SUMMARY:
The purpose of this study is to see if a new Smart Phone application can help Veterans manage their panic symptoms after completing a two-day treatment for panic attacks.

DETAILED DESCRIPTION:
The first goal is to see how helpful the Smart Phone application is in helping veterans with panic symptoms continue to improve after you complete treatment.

The second goal of this study is to find out how much veterans like the Smart Phone application.

The third goal is to see how practical it is to use the Smart Phone application as a form of follow-up care. We want to see how much time is needed to provide technical support in using the application.

ELIGIBILITY:
Inclusion Criteria:

Participants must

1. be an Operation Enduring Freedom/Operation Iraqi Freedom/Operation New Dawn (OEF/OIF/OND) Veteran
2. currently meet criteria for PD with or without Agoraphobia
3. complete the weekend PD treatment at the Lufkin, Conroe or Texas City CBOC.

Exclusion Criteria:

1. current substance dependence
2. organic psychosis
3. symptomatic bipolar disorder
4. severe depression with suicidal intent or plan
5. cognitive impairment (indicated by scores <20 on SLUMS)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2011-04; Primary Completion 2013-05 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Panic Control Treatment (PCT) | 2 days
  A cognitive-behavioral therapy for PD that is highly efficacious, the standard delivery format of these sessions are typically offered once a week over a period of several months. This can pose challenges to rural Veterans who have multiple commitments and face long travel distances for mental health services.
  To improve accessibility to panic treatment, one innovative approach has been to deliver PCT in an intensive, two-day format.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Teng, Ph.D, Principal Investigator — Michael E. DeBakey VA Medical Center
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, Texas, United States